CLINICAL TRIAL: NCT07301827
Title: Study on the Diagnostic Value of Novel PET Molecular Imaging for Renal Cell Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: XLan-0923
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Renal Cell Carcinoma
Keywords: Renal cell carcinoma; PET imaging; PSMA; CAIX; CD70
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — gallium 68 PSMA-11

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PET imaging targeting CAIX in renal cell carcinoma (Experimental)
  Interventions: Drug: [68Ga]Ga-DOTA-CAIX peptide
- PET imaging targeting PSMA in renal cell carcinoma (Experimental)
  Interventions: Drug: [68Ga]Ga-PSMA
- PET imaging targeting CD70 in renal cell carcinoma (Experimental)
  Interventions: Drug: [68Ga]Ga-NOTA-CD70 antibody fragment

INTERVENTIONS:
Drug: [68Ga]Ga-DOTA-CAIX peptide — To perform integrated PET/MR or PET/CT visualization of patients with clinically suspected or confirmed renal cell carcinoma with high CAIX expression and healthy volunteers, using specific positron imaging agents targeting CAIX (taking [68Ga]Ga-DOTA-CAIX peptide as an example), to achieve the following purposes: Patients with malignant tumors: for diagnosis and staging of diseases, comparing with the gold standard pathological diagnosis, evaluating diagnostic efficacy, clarifying the presence or absence of lesions, and determining the location and nature of lesions; comparing with [18F]FDG PET for accurate staging, evaluating the tumor load, and helping to determine the therapeutic plan.
  Healthy volunteers: Pharmacokinetic analysis will be performed to clarify the distribution and metabolism of the drug in the body and its safety.
  Arms: PET imaging targeting CAIX in renal cell carcinoma
Drug: [68Ga]Ga-NOTA-CD70 antibody fragment — To perform integrated PET/MR or PET/CT visualization of patients with clinically suspected or confirmed renal cell carcinoma with high CD70 expression and healthy volunteers, using specific positron imaging agents targeting CD70 (taking [68Ga]Ga-NOTA-CD70 antibody fragment as an example), to achieve the following purposes: Patients with malignant tumors: for diagnosis and staging of diseases, comparing with the gold standard pathological diagnosis, evaluating diagnostic efficacy, clarifying the presence or absence of lesions, and determining the location and nature of lesions; comparing with [18F]FDG PET for accurate staging, evaluating the tumor load, and helping to determine the therapeutic plan.
  Arms: PET imaging targeting CD70 in renal cell carcinoma
Drug: [68Ga]Ga-PSMA — To perform integrated PET/MR or PET/CT visualization of patients with clinically suspected or confirmed renal cell carcinoma with high PSMA expression and healthy volunteers, using specific positron imaging agents targeting PSMA (taking [68Ga]Ga-PSMA as an example), to achieve the following purposes: Patients with malignant tumors: for diagnosis and staging of diseases, comparing with the gold standard pathological diagnosis, evaluating diagnostic efficacy, clarifying the presence or absence of lesions, and determining the location and nature of lesions; comparing with [18F]FDG PET for accurate staging, evaluating the tumor load, and helping to determine the therapeutic plan.
  Arms: PET imaging targeting PSMA in renal cell carcinoma

SUMMARY:
This study is a diagnostic study. This project aims to explore the clinical application value of PET imaging technologies targeting PSMA, CAIX, and CD70 in renal cell carcinoma. By utilizing PSMA-targeted PET radiopharmaceuticals (e.g., [⁶⁸Ga]Ga-PSMA), CAIX-targeted PET radiopharmaceuticals (e.g., [⁶⁸Ga]Ga-DOTA-CAIX), and CD70-targeted PET radiopharmaceuticals (e.g., [⁶⁸Ga]Ga-NOTA-CD70 antibody fragment) in patients with clinically suspected or confirmed renal cell carcinoma and healthy volunteers, we will investigate their diagnostic and therapeutic potential. [⁶⁸Ga]Ga-DOTA-CAIX peptide as an example), and a PET imaging agent targeting CD70 ([⁶⁸Ga]Ga-NOTA-CD70 antibody fragment as an example) in patients with clinically suspected or confirmed renal cell carcinoma and healthy volunteers. Integrated PET/MR or PET/CT imaging will be performed to aid in the diagnosis and staging of renal cell carcinoma, assess tumor burden and the expression levels of PSMA, CAIX, and CD70, and assist in determining treatment strategies. Concurrently, preliminary pharmacokinetic analysis of the novel CAIX-targeting molecular probe will be conducted in healthy volunteers to elucidate its metabolic patterns and adverse reactions in vivo.

DETAILED DESCRIPTION:
Malignant tumors represent one of the major diseases threatening human health, with their incidence and mortality rates continuing to rise and showing a trend toward younger age groups, presenting a severe challenge for prevention and treatment. Renal cell carcinoma (RCC) is the most common pathological type among kidney malignancies, accounting for approximately 70% of all kidney cancers. As a highly invasive tumor, approximately 30% of RCC patients present with distant metastases at initial diagnosis, and the postoperative recurrence or metastasis rate also reaches 30%. Therefore, early precise diagnosis and accurate tumor burden assessment are crucial for improving patient prognosis, and rational clinical staging forms the foundation for developing individualized treatment strategies.

Currently, imaging diagnosis and postoperative monitoring of renal cell carcinoma primarily rely on contrast-enhanced computed tomography (CT), but this method has limitations, particularly the lack of efficient and reliable whole-body assessment tools. Due to the generally low uptake of 18F-fluorodeoxyglucose ([18F]FDG) in RCC, the application value of conventional [18F]FDG positron emission tomography/computed tomography (PET/CT) in RCC diagnosis and monitoring is limited. Furthermore, [18F]FDG PET/CT lacks sufficient specificity in distinguishing benign from malignant renal masses, as some benign lesions may also exhibit increased FDG uptake. Consequently, developing highly sensitive and specific molecular imaging methods to optimize RCC diagnosis and staging has become an urgent clinical priority.

Nuclear medicine testing targeting RCC-specific markers holds promise for addressing this challenge. In recent years, prostate-specific membrane antigen (PSMA) PET/CT imaging has demonstrated significant value in prostate cancer staging. Multiple studies indicate PSMA overexpression in endothelial cells of neovascularization across various tumors. Although preliminary data suggest PSMA PET/CT may aid in predicting RCC histological grading and adverse prognosis, its precise role in RCC clinical management remains unclear. Furthermore, based on multi-omics analysis and large-scale pathological studies, carbonic anhydrase IX (CAIX) and CD70 have been identified as two prominent potential specific targets in RCC.

CAIX, a transmembrane metalloproteinase involved in regulating tumor microenvironment pH, exhibits a significant positive correlation between its expression levels and tumor hypoxia, making it an important marker for poor prognosis. Notably, due to VHL gene inactivation mutations and subsequent sustained activation of the downstream HIF-1α signaling pathway, CAIX expression is upregulated in over 95% of RCC cases. Beyond the gastrointestinal and biliary tract systems, CAIX is scarcely detectable in normal tissues, making it an ideal target for molecular imaging and targeted therapy in RCC.

CD70 (CD27 ligand), belonging to the tumor necrosis factor superfamily (TNFSF7), is normally expressed transiently on activated T cells, B cells, NK cells, and mature dendritic cells under physiological conditions. Recent studies indicate that CD70 is abnormally overexpressed in 78% of clear cell RCC and 32% of papillary RCC, while absent in normal renal tissue. Furthermore, dysregulation of the CD70-CD27 axis in tumor cells and the microenvironment contributes to immune evasion and tumor progression. CD70 expression on tumor cells is also strongly associated with poor prognosis in multiple malignancies. Currently, eliminating CD70-positive tumor cells or blocking the CD70-CD27 signaling axis represents a novel therapeutic direction for renal cell carcinoma. Monoclonal antibodies and antibody-drug conjugates targeting CD70 have entered clinical trial phases. Therefore, developing a radiolabeled tracer targeting CD70 holds significant clinical and practical value. It not only facilitates precise diagnosis and staging of RCC but also provides crucial evidence for studying CD70-related immunotherapy mechanisms.

In summary, this project aims to explore the clinical application value of PET imaging technologies targeting PSMA, CAIX, and CD70 in renal cell carcinoma. By utilizing PSMA-targeted PET radiopharmaceuticals (e.g., [68Ga]Ga-PSMA), CAIX-targeted PET tracers (e.g., [68Ga]Ga-DOTA-CAIX peptide), and CD70-targeted PET tracers (e.g., [68Ga]Ga-NOTA-CD70 antibody fragment) in clinically suspected or confirmed renal cell carcinoma patients and healthy volunteers. Integrated PET/MR or PET/CT imaging will be performed to facilitate diagnosis and staging of renal cell carcinoma, assess tumor burden, and evaluate PSMA and CD70 expression, assisting in determining treatment strategies. Concurrently, preliminary pharmacokinetic analysis of the novel CAIX-targeting molecular probe will be conducted in healthy volunteers to elucidate its metabolic patterns and adverse reactions in vivo.

ELIGIBILITY:
Inclusion Criteria:

Tumor subjects:

1. The subject or his/her legal representative is able to sign the informed consent form signed and dated;
2. Promise to abide by the research procedures and cooperate with the implementation of the whole process of research;
3. Adult subjects (aged 18 years or above), male or female;
4. Patients with clinically suspected or confirmed renal cell carcinoma (supporting evidence includes serum-related tumor markers, ultrasound, CT, MRI and other imaging data and histopathological examinations, etc.), and are in good general condition;
5. Conform to specific laboratory test results;
6. Contraception for at least one month before screening for females in the childbearing period, and commitment to use contraception throughout the study period and continue until the specified time after the end of the study;
7. Other set selection criteria.

Healthy Subjects:

1. Fully understand and voluntarily sign the informed consent form;
2. Male or female, age 18-70 years old;
3. Male weight >=50.0kg, female weight >=45.0kg; Body mass index (BMI) within the range of 19.0~26.0kg/m^2 (including the cut-off value);
4. No history of chronic or serious diseases such as cardiovascular, liver, kidney, respiratory, blood and lymphatic, endocrine, immunologic, psychiatric, neuromuscular, gastrointestinal system, etc., within three years, and in good general health;
5. There is no abnormality in vital signs examination and physical examination;
6. Have no fertility plan during the trial and within 6 months after the end of the trial and voluntarily take effective contraceptive measures and have no sperm and egg donation plans;
7. Able to communicate well with the investigator, and understand and comply with the requirements of the study.

Exclusion Criteria:

Tumor subjects:

1. Those who are unable to complete PET/MR or PET/CT examination (including inability to lie flat, claustrophobia, radiophobia, etc.);
2. Patients with known hypersensitivity to targeted PSMA, CAIX or CD70 PET imaging agents or synthetic excipients; The fasting blood glucose level before injection of [18F]FDG exceeded 11.0 mmol/L;
3. Patients who are pregnant or lactating;
4. Those who have other factors that are not suitable for participating in this test.

Healthy Subjects:

1. Any serious or unstable medical condition; Those who have acute illness before the study; Previous or existing malignancy;
2. Pregnant and lactating women;
3. Those who have undergone surgery within 6 months before the trial, which is judged by the investigator to affect absorption, distribution, metabolism, and excretion;
4. Those who have used any drugs (including prescription drugs, over-the-counter drugs, and Chinese herbal medicines) within 2 weeks before the trial;
5. Participation in other research studies involving radioactive materials (within the past 12 months);
6. Any other factors that affect the results of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Visual and standardized uptake values assessment of lesions and biodistribution | 1 year
  At least two experienced nuclear medicine physicians will conduct a visual analysis using consensus reading. The standardized uptake value (SUV) of tumor and organs will be measured after a semiquantitative analysis is conducted for each case. The SUV ranges from 0 to infinity, and a higher score means a higher uptake of nuclear probe by the tumor, which implies a greater threat of the tumor being malignant or higher stage.

SECONDARY OUTCOMES:
Radioactivity in the blood and urine samples | Blood samples were collected at 25 minutes, 55 minutes and 115 minutes after injection.
Pathological sections of tumor tissue | up to 1 year
  The excised tumour tissue was taken for immunohistochemistry to verify its target expression

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No